CLINICAL TRIAL: NCT02974595
Title: Studies of the Natural History, Pathogenesis, and Outcome of Autoinflammatory Diseases (NOMID/CAPS, DIRA, CANDLE, SAVI, NLRC4-MAS, Still'S-like Diseases, and Other Undifferentiated Autoinflammatory Diseases)
Brief Title: Natural History, Pathogenesis, and Outcome of Autoinflammatory Diseases (NOMID/CAPS, DIRA, CANDLE, SAVI, NLRC4-MAS, Still'S-like Diseases, and Other Undifferentiated Autoinflammatory Diseases)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170016; 17-I-0016
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01-07

CONDITIONS: NOMID; DIRA; NLRC4-MAS; SAVI; CANDLE
Keywords: Study of pathogenesis of patients affected with autoinflammatory diseases; This Includes the Clinical, Immunological , Genetic, and Metabolic Characteristi; Collection of Clinical and Laboratory Outcome Data; Evaluation of Characteristics/Disease Manifestations; Natural History
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Affected Participants: Individuals with undifferentiated autoinflammatory diseases or genetically defined conditions, such as NOMID/CAPS, DIRA, CANDLE, SAVI, and NLRC4 MAS.
- Healthy Volunteer: Volunteers without known autoinflammatory disease who consent to providing blood specimen for genetic testing.
- Unaffected Relatives: Blood relatives of the affected patients without known autoinflammatory disease who consent to providing specimen for genetic testing.

SUMMARY:
Background:

Some diseases cause chronic inflammation with intermittent flares in the body. These are called autoinflammatory diseases. They can cause fevers, rashes, ulcers, and other problems. Researchers want to learn more about the causes and effects of these diseases. They hope this will improve how the disease is managed in the future.

Objectives:

To understand the underlying immune dysregulation

To identify the genetic cause

To translate our findings into novel treatments that improve patients disease outcomes

Eligibility:

Patients with known NOMID/CAPS, DIRA, CANDLE, SAVI, NLRC4-MAS, Still's Disease, and with other yet undifferentiated autoinflammatory diseases.

Unaffected relatives of participants with a known or undifferentiated autoinflammatory disease

Healthy adult volunteers at least 18 years of age

Design:

Participants will be screened with blood sample and medical history. They may provide copies of their medical records.

Enrolled participants will be evaluated at the NIH for 2-5 days. All participants will have a detailed medical history, physical exam, blood tests, and other evaluations depending on the extent of their autoinflammatory disease.

Participants may also expect the following assessments:

1. Clinical tests that help assess organ damage and function such as hearing, vision, memory, and learning tests.
2. Imaging studies to characterize organ involvement of the inflammatory disease including: X-rays, CT scans, special MRIs, and bone scans.
3. Laboratory evaluations including clinical markers of disease activity, research samples for genetic studies, blood samples for cytokine/biomarker assessment, and gene expression profiling.
4. Questionnaires to assess disease activity and quality of life.
5. If indicated, other procedures may be administered that include: a lumbar puncture if CNS inflammation is suspected, a skin biopsy if skin inflammation is present, and/or gastrointestinal and pulmonary procedures if they are clinically indicated.

Participants may return for a single follow-up visit or for long-term follow-up visits depending on their disease and willingness to return. Long-term follow-up may occur for up to 15 years on this protocol.

DETAILED DESCRIPTION:
Autoinflammatory diseases are a group of immune dysregulatory diseases that are characterized by recurrent episodes of systemic as well as organ-specific inflammation that can involve the skin, eyes, joints, bones, muscles, lungs, serosal surfaces, inner ear, brain, and other organs. The prominent role of IL-1 in the pathogenesis of these disorders first became evident through the discovery of mutations in the gene NLRP3 and IL1RN. Since then, we have identified additional mutations that cause autoinflammatory diseases, including mutations in proteasome components and STING1 that suggest a role of increased type I IFN signaling as a contributor to the disease pathogenesis of autoinflammatory diseases and in NLRC4 and CDC42 that suggest a role of IL-18 in some autoinflammatory diseases. In this natural history study, we seek to comprehensively evaluate people with autoinflammatory diseases that include clinical, genetic, immunologic, andendocrinologic characterizations. Other rare diseases not mediated by IL-1, IL-18 or type I IFN and presumed to be autoinflammatory diseases with unknown genetic causes may also be eligible under this protocol. In addition, we intend to evaluate long-term outcomes and biomarkers over time in selected diseases. We plan to follow most participants for the duration of this study (15 years). Relatives who do not have autoinflammatory diseases as well as healthy volunteers will also be recruited to serve as controls for biomarker, genetic, and other molecular analyses.

ELIGIBILITY:
* INCLUSION CRITERIA - AFFECTED PARTICIPANTS:

  1. Be 2 to 99 years old for participants who will be seen at the NIH CC; be 0 (newborn) to 99 years old for participants who participate remotely via a virtual protocol visit and will submit mail-in samples. Participants younger than 3 years will be seen in the outpatient clinic at the NIH CC if approved by the Pediatric

     Consult Service as per NIH CC policy and guidelines.
  2. Is willing to allow storage of biological specimens for future use in medical research.
  3. Is willing to allow genetic testing on collected biological samples.
  4. Has a primary care or other physician who will manage all health conditions related or unrelated to the study objectives.
  5. Fulfills one of the following criteria:

     * Has a known disease-causing genetic mutation associated with NOMID/CAPS, DIRA, CANDLE, SAVI, or NLRC4-MAS.
     * Has clinical signs or symptoms not explained by any other disorder (eg, infections, malignancies) and are consistent with a possible IL-1 mediated autoinflammatory disease. Participants must meet both of the following criteria:

       * Clinical characteristics strongly consistent with an IL-1 mediated autoinflammatory disease per the following criteria and at the discretion of the principal investigator (PI). Individuals must have a past or present history of one of the following to be considered for study enrollment:

         * Recurrent fever that has gone undiagnosed after reasonable attempts, and that is consistent with the conditions under study in this protocol
         * Neutrophilic urticaria, pustular dermatitis, erysipelas-like erythema, or urticarial rash
         * Epiphyseal and/or patella enlargement, periostitis, myalgias, arthralgias, arthritis, or recurrent multifocal aseptic osteomyelitis
         * Sensorineural hearing loss
         * Chronic aseptic meningitis or CNS vasculitis
         * Conjunctivitis, episcleritis, uveitis, papilledema, pleuritis, pericarditis, aseptic peritonitis, early onset enterocolitis, hepatosplenomegaly, or lymphadenopathies
       * Laboratory characteristics strongly consistent with an IL-1mediated autoinflammatory disease per the following criteria. Individuals must havepast or present history of evidence of systemic inflammation (eg, elevation of C-reactive protein [CRP] and/or erythrocyte sedimentation rate [ESR], anemia, thrombocytosis).
     * Has clinical signs or symptoms not explained by any other disorder (eg, infections, malignancies) and are consistent with a possible IFN-mediated, autoinflammatory disease.1,36 Participants must meet both of the following criteria:

       * Clinical characteristics strongly consistent with an IFN-mediated autoinflammatory disease per the following criteria and at the discretion of the PI. Individuals must have a past or present history of one of the following to be considered for study enrollment:

         * Recurrent fevers that has gone undiagnosed after reasonable attempts, and that is consistent with the conditions under study in this protocol
         * Panniculitis, ischemic ulcerative skin lesions, chilblain lesions, or livedo reticularis
         * Lipodystrophy
         * Myositis, arthralgias, arthritis, or joint contractures
         * Basal ganglia calcifications or white matter CNS disease
         * Interstitial lung disease, lung fibrosis, or pulmonary hypertension
         * Conjunctivitis, episcleritis, cortical blindness, glaucoma, papilledema, or hepatosplenomegaly
         * Laboratory characteristics strongly consistent with an IFN-mediated autoinflammatory disease per the following criteria. Individuals must have past or present history one or more of the following to be considered for study enrollment:
         * Evidence of systemic inflammation (eg, ESR or CRP)
         * Cytopenias (eg. leukopenia, anemia, or thrombocytopenia)
         * Dyslipidemia or insulin resistance
         * Abnormal liver function test, creatinine kinase (CK), or LDH
     * Has clinical signs or symptoms consistent with an undifferentiated autoinflammatory disease (including but not limited to dysregulation in other proinflammatory cytokines such as IL-17, TNF, IL-18, and others). Participants must meet one of the following criteria:

       * Clinical characteristics strongly consistent with an undifferentiated autoinflammatory disease. Individuals must have a past or present history of one of the clinical and one of the laboratory characteristics mentioned above to be considered for study enrollment.
       * Individuals with defined organ inflammation associated with past or current evidence of systemic inflammation.
  6. Alternatively to #5, had been enrolled in the past as an affected participant on NIAMS study 03-AR-0173 and or had samples collected on 03-AR-0173.

INCLUSION CRITERIA - UNAFFECTED RELATIVES OF AFFECTED PARTICIPANTS:

1. Be 2 to 99 years old for participants who will be seen at the NIH CC; be 0 (newborn) to 99 years old for participants who participate remotely via a virtual protocol visit and will submit mail-in samples. Participants younger than 3 years will be seen in the outpatient clinic at the NIH CC if approved by the Pediatric Consult Service as per NIH CC policy and guidelines.)
2. Be related by blood to an affected participant.
3. Is willing to allow storage of biological samples for future use in medical research.
4. Is willing to allow genetic testing on collected biological samples.
5. Does not fulfill any of inclusion criterion #5 for affected participants.
6. Is able to provide informed consent.

INCLUSION CRITERIA - HEALTHY VOLUNTEERS:

1. Be at least 18 years old.
2. Not be related to an affected participant.
3. s willing to allow storage of biological samples for future use in medical research.
4. Is willing to allow genetic testing on collected biological samples.
5. Does not fulfill any of inclusion criterion #5 for affected participants.
6. Is able to provide informed consent.

PARTICIPANT EXCLUSION CRITERIA:

1. Presence of conditions that, in the judgment of the investigator, may put the participant at undue risk or make them unsuitable for participation in the study.
2. Oncological evaluation suggestive of lymphoma, leukemia or multiple myeloma, except for participants with a known primary diagnosis of an autoinflammatory disease who subsequently developed a malignancy. These patients will not be excluded from the study.

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population is quite diverse as affected participants are from all over the world, different age ranges, and all race/ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2016-12-09 (Actual); Primary Completion 2031-08-31 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
To study the pathogenesis of patients affected with auto-inflammatory diseases, including their clinical, immunological, genetic and metabolic/endocrinological characteristics. | 1-2 years, 3-5 years, 10 years
  To study the pathogenesis of patients affected with autoinflammatory diseases, including their clinical, immunological, genetic and metabolic/endocrinological characteristics.

SECONDARY OUTCOMES:
Longitudinal fluctuations in clinical and biomarker characteristics of autoinflammatory diseases | 1-2 years, 3-5 years, 10 years
  To evaluate clinical characteristics/disease manifestations and blood, body fluids, and tissue biomarkers during disease flares and quiescence.
Long term Organ specific outcome (clinical and biomarker evidence of both inflammation and damage accrual) | 1-2 years, 3-5 years, 10 years
  To collect long-term clinical and laboratory outcome parameters of the multiorgan inflammatory involvement and/or organ damage in patients with genetically defined or undifferentiated autoinflammatory (immune-dysregulatory) diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Raphaela T Goldbach-Mansky, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
As outlined in our approved GDS Plan (dated 09/27/2019): Whole exome and whole genome sequencing data
Supporting Information: Study Protocol
Time Frame: As outlined in our approved GDS Plan (dated 09/27/2019) and protocol: Following genetic testing, the data will be shared in a controlled-access public database for other investigators to benefit from it (eg, dbGaP, the Database of Genotypes and Phenotypes).
Access Criteria: Other NIH and non-NIH investigators may use these data/specimens for research purposes. @@@IRB review and approval will be obtained for all research involving identifiable data/specimen, including any coded and linked samples or data that can be linked back to the respective subjects.@@@@@@We will share human data generated in this study for future research through:@@@Our NIH-funded and approved public repository for genetic and RNA sequence data: De-identified data will be shared per our approved Genetic Data Sharing Plan. @@@BTRIS (Biomedical Translational Research Information System) sharing activities in the NIH Clinical Center (CC): includes Identifiable data generated in CC. @@@Appropriate individual regulatory approvals will govern sharing of data/specimens with outside collaborators.@@@Data will be shared with medical professionals involved in clinical care of each patient to assist with medical care of the patient. @@@Publication and/or public presentations. @@@

REFERENCES:
- [Background] Bhuyan F, de Jesus AA, Mitchell J, Leikina E, VanTries R, Herzog R, Onel KB, Oler A, Montealegre Sanchez GA, Johnson KA, Bichell L, Marrero B, De Castro LF, Huang Y, Calvo KR, Collins MT, Ganesan S, Chernomordik LV, Ferguson PJ, Goldbach-Mansky R. Novel Majeed Syndrome-Causing LPIN2 Mutations Link Bone Inflammation to Inflammatory M2 Macrophages and Accelerated Osteoclastogenesis. Arthritis Rheumatol. 2021 Jun;73(6):1021-1032. doi: 10.1002/art.41624. Epub 2021 May 9. PMID 33314777
- [Background] Goldbach-Mansky R, Dailey NJ, Canna SW, Gelabert A, Jones J, Rubin BI, Kim HJ, Brewer C, Zalewski C, Wiggs E, Hill S, Turner ML, Karp BI, Aksentijevich I, Pucino F, Penzak SR, Haverkamp MH, Stein L, Adams BS, Moore TL, Fuhlbrigge RC, Shaham B, Jarvis JN, O'Neil K, Vehe RK, Beitz LO, Gardner G, Hannan WP, Warren RW, Horn W, Cole JL, Paul SM, Hawkins PN, Pham TH, Snyder C, Wesley RA, Hoffmann SC, Holland SM, Butman JA, Kastner DL. Neonatal-onset multisystem inflammatory disease responsive to interleukin-1beta inhibition. N Engl J Med. 2006 Aug 10;355(6):581-92. doi: 10.1056/NEJMoa055137. PMID 16899778
- [Background] Liu Y, Ramot Y, Torrelo A, Paller AS, Si N, Babay S, Kim PW, Sheikh A, Lee CC, Chen Y, Vera A, Zhang X, Goldbach-Mansky R, Zlotogorski A. Mutations in proteasome subunit beta type 8 cause chronic atypical neutrophilic dermatosis with lipodystrophy and elevated temperature with evidence of genetic and phenotypic heterogeneity. Arthritis Rheum. 2012 Mar;64(3):895-907. doi: 10.1002/art.33368. PMID 21953331
- [Background] Liu Y, Jesus AA, Marrero B, Yang D, Ramsey SE, Sanchez GAM, Tenbrock K, Wittkowski H, Jones OY, Kuehn HS, Lee CR, DiMattia MA, Cowen EW, Gonzalez B, Palmer I, DiGiovanna JJ, Biancotto A, Kim H, Tsai WL, Trier AM, Huang Y, Stone DL, Hill S, Kim HJ, St Hilaire C, Gurprasad S, Plass N, Chapelle D, Horkayne-Szakaly I, Foell D, Barysenka A, Candotti F, Holland SM, Hughes JD, Mehmet H, Issekutz AC, Raffeld M, McElwee J, Fontana JR, Minniti CP, Moir S, Kastner DL, Gadina M, Steven AC, Wingfield PT, Brooks SR, Rosenzweig SD, Fleisher TA, Deng Z, Boehm M, Paller AS, Goldbach-Mansky R. Activated STING in a vascular and pulmonary syndrome. N Engl J Med. 2014 Aug 7;371(6):507-518. doi: 10.1056/NEJMoa1312625. Epub 2014 Jul 16. PMID 25029335
- [Derived] Lee Y, Wessel AW, Xu J, Reinke JG, Lee E, Kim SM, Hsu AP, Zilberman-Rudenko J, Cao S, Enos C, Brooks SR, Deng Z, Lin B, de Jesus AA, Hupalo DN, Piotto DG, Terreri MT, Dimitriades VR, Dalgard CL, Holland SM, Goldbach-Mansky R, Siegel RM, Hanson EP. Genetically programmed alternative splicing of NEMO mediates an autoinflammatory disease phenotype. J Clin Invest. 2022 Mar 15;132(6):e128808. doi: 10.1172/JCI128808. PMID 35289316
- [Derived] Kim H, Gunter-Rahman F, McGrath JA, Lee E, de Jesus AA, Targoff IN, Huang Y, O'Hanlon TP, Tsai WL, Gadina M, Miller FW, Goldbach-Mansky R, Rider LG. Expression of interferon-regulated genes in juvenile dermatomyositis versus Mendelian autoinflammatory interferonopathies. Arthritis Res Ther. 2020 Apr 6;22(1):69. doi: 10.1186/s13075-020-02160-9. PMID 32252809
- [Derived] de Jesus AA, Hou Y, Brooks S, Malle L, Biancotto A, Huang Y, Calvo KR, Marrero B, Moir S, Oler AJ, Deng Z, Montealegre Sanchez GA, Ahmed A, Allenspach E, Arabshahi B, Behrens E, Benseler S, Bezrodnik L, Bout-Tabaku S, Brescia AC, Brown D, Burnham JM, Caldirola MS, Carrasco R, Chan AY, Cimaz R, Dancey P, Dare J, DeGuzman M, Dimitriades V, Ferguson I, Ferguson P, Finn L, Gattorno M, Grom AA, Hanson EP, Hashkes PJ, Hedrich CM, Herzog R, Horneff G, Jerath R, Kessler E, Kim H, Kingsbury DJ, Laxer RM, Lee PY, Lee-Kirsch MA, Lewandowski L, Li S, Lilleby V, Mammadova V, Moorthy LN, Nasrullayeva G, O'Neil KM, Onel K, Ozen S, Pan N, Pillet P, Piotto DG, Punaro MG, Reiff A, Reinhardt A, Rider LG, Rivas-Chacon R, Ronis T, Rosen-Wolff A, Roth J, Ruth NM, Rygg M, Schmeling H, Schulert G, Scott C, Seminario G, Shulman A, Sivaraman V, Son MB, Stepanovskiy Y, Stringer E, Taber S, Terreri MT, Tifft C, Torgerson T, Tosi L, Van Royen-Kerkhof A, Wampler Muskardin T, Canna SW, Goldbach-Mansky R. Distinct interferon signatures and cytokine patterns define additional systemic autoinflammatory diseases. J Clin Invest. 2020 Apr 1;130(4):1669-1682. doi: 10.1172/JCI129301. PMID 31874111
- [Derived] Sanchez GAM, Reinhardt A, Ramsey S, Wittkowski H, Hashkes PJ, Berkun Y, Schalm S, Murias S, Dare JA, Brown D, Stone DL, Gao L, Klausmeier T, Foell D, de Jesus AA, Chapelle DC, Kim H, Dill S, Colbert RA, Failla L, Kost B, O'Brien M, Reynolds JC, Folio LR, Calvo KR, Paul SM, Weir N, Brofferio A, Soldatos A, Biancotto A, Cowen EW, Digiovanna JJ, Gadina M, Lipton AJ, Hadigan C, Holland SM, Fontana J, Alawad AS, Brown RJ, Rother KI, Heller T, Brooks KM, Kumar P, Brooks SR, Waldman M, Singh HK, Nickeleit V, Silk M, Prakash A, Janes JM, Ozen S, Wakim PG, Brogan PA, Macias WL, Goldbach-Mansky R. JAK1/2 inhibition with baricitinib in the treatment of autoinflammatory interferonopathies. J Clin Invest. 2018 Jul 2;128(7):3041-3052. doi: 10.1172/JCI98814. Epub 2018 Jun 11. PMID 29649002
- [Derived] Kim H, de Jesus AA, Brooks SR, Liu Y, Huang Y, VanTries R, Montealegre Sanchez GA, Rotman Y, Gadina M, Goldbach-Mansky R. Development of a Validated Interferon Score Using NanoString Technology. J Interferon Cytokine Res. 2018 Apr;38(4):171-185. doi: 10.1089/jir.2017.0127. PMID 29638206
- [Derived] Kim H, Brooks KM, Tang CC, Wakim P, Blake M, Brooks SR, Montealegre Sanchez GA, de Jesus AA, Huang Y, Tsai WL, Gadina M, Prakash A, Janes JM, Zhang X, Macias WL, Kumar P, Goldbach-Mansky R. Pharmacokinetics, Pharmacodynamics, and Proposed Dosing of the Oral JAK1 and JAK2 Inhibitor Baricitinib in Pediatric and Young Adult CANDLE and SAVI Patients. Clin Pharmacol Ther. 2018 Aug;104(2):364-373. doi: 10.1002/cpt.936. Epub 2017 Dec 8. PMID 29134648
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-I-0016.html